CLINICAL TRIAL: NCT06421493
Title: Role of the Maternal Microbiota on the Immune Response and Metabolism During Hypertensive Disorders
Acronym: MATER
Status: Recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 0004622
Record Dates: First submitted 2024-05-07; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Preeclampsia
Keywords: microbiome; immune system; metabolome
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The protocol involves analyzing the maternal microbiota and metabolome from fecal samples and blood samples collected from women who have consented to the study.
  The blood will be centrifuged to separate the plasma from the cellular fraction. The isolated plasma will be frozen at -80°C for subsequent metabolomic and microbiota analyses, while the cells will be resuspended in phosphate-buffered saline (PBS) in equal volume to the isolated plasma. focal material will be stored at -80°C.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Age > 18 years Singleton pregnancy Live fetus at 11-13 weeks of gestation Pregnancies complicated by hypertensive disorders (HDP) and fetal growth restriction (FGR) Women with pregnancies complicated by HDP and a fetus with appropriate weight for gestational age (AGAf) Women with pregnancies complicated solely by early fetal growth restriction (before 34 weeks) Women with pregnancies complicated solely by late fetal growth restriction (after 34 weeks) Women identified as high-risk in first-trimester screening for preeclampsia Women identified as high-risk in first-trimester screening for fetal growth restriction
- Controls: Age > 18 years Singleton pregnancy Feto vivo a 11-13 settimane di gravidanza Low-risk pregnancies in first-trimester screening for preeclampsia and fetal growth restriction, with physiological follow-up visits until delivery (homogeneous control sample)

SUMMARY:
Preeclampsia (PE) is a significant cause of maternal and fetal morbidity and mortality, characterized by high blood pressure and proteinuria during pregnancy. It has two main phenotypes: one linked to placental damage and the other to metabolic factors like obesity. Early identification of high-risk groups is crucial, though there's ongoing disagreement over its classification. Research suggests a potential connection between maternal gut bacteria and PE, offering avenues for improved prevention strategies. This study aims to investigate the differences in maternal gut microbiota between these two PE phenotypes.

DETAILED DESCRIPTION:
Preeclampsia (PE) is one of the leading causes of maternal and fetal morbidity and mortality. It is defined as the presence of systolic blood pressure (SBP) ≥ 140 and diastolic blood pressure (DBP) ≥ 90 on two consecutive measurements six hours apart, associated with proteinuria >300 mg/24 h or 2++ detected by urine dipstick or the presence of organ damage or intrauterine growth restriction. Preeclampsia complicates 3-8% of pregnancies and is responsible for more than 76,000 maternal deaths annually.

Scientific evidence suggests the existence of two distinct phenotypes of the disease: preeclampsia due to placental damage and preeclampsia on a metabolic basis. The former phenotype recognizes altered invasion of the maternal endometrium by the trophoblast as its pathogenesis, where defective trophoblast invasion leads to the development of preeclampsia often associated with early presentation in pregnancy, intrauterine growth restriction (IUGR), and the need for delivery at low gestational ages. The latter phenotype recognizes a metabolic basis, which represents about 4% of hypertensive disorders of pregnancy (HDP), and is dependent on maternal predisposition in patients with visceral obesity and metabolic syndrome.

Evidence suggests that maternal risk factors for metabolic dysfunction may lead to late placental dysfunction in pregnancy. Metabolic-based preeclampsia manifests in patients with pre-existing low-grade inflammation related to truncal obesity and metabolic syndrome, compounded by pregnancy-related inflammation and insulin resistance.

Today, starting as early as the first trimester of pregnancy, maternal cardiovascular and hemodynamic function can be assessed using a non-invasive and safe method for both the mother and fetus through the USCOM (Ultra Sonic Cardiac Output Monitor) system. This system provides real-time data on numerous central and peripheral hemodynamic parameters.

There is still disagreement among scientific societies regarding the classification of preeclampsia and its possible different clinical phenotypes, making personalized clinical approaches to this condition challenging. However, early identification of high-risk groups is becoming increasingly important for diagnostic follow-up and therapeutic strategies based on pathogenesis.

Recently, a screening method at 11-13 weeks of gestation has been developed to predict 75% of pregnancies that will develop preterm preeclampsia (<37 weeks of gestation) based on a risk calculation algorithm combining weight and height measurements, mean arterial pressure measured with automated devices, blood sampling for PLGF measurement, and Doppler ultrasound measurement of the mean pulsatility index (PI) of the uterine arteries.

However, this screening method can only predict a portion of patients who will develop preeclampsia before 37 weeks and who may benefit from aspirin intake if administered at doses >100mg and before 16 weeks. Predicting and effectively preventing preeclampsia that occurs after 37 weeks remains the subject of debate and scientific research.

Among emerging etiopathogenetic hypotheses, numerous scientific publications suggest that alterations in maternal immunity and immune tolerance are the basis of hypertensive disorders in pregnancy. Recent discoveries suggest that changes in maternal intestinal microbiota may underlie these immune alterations. Alterations in gut microbiota diversity and composition, known as "dysbiosis," can influence systemic immune responses and metabolic disturbances such as gestational diabetes and preeclampsia, posing risks of metabolic alterations in the neonate.

Based on these premises, this study aims to define the characteristics of maternal intestinal microbiota in the two different clinical phenotypes of preeclampsia: placental preeclampsia associated with growth restriction and metabolic-based preeclampsia associated with a fetus of appropriate weight for gestational age.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Singleton pregnancy
* Live fetus at 11-13 weeks of gestation
* Pregnancies complicated by hypertensive disorders (HDP) and fetal growth restriction (FGR) Women with pregnancies complicated by HDP and a fetus with appropriate weight for gestational age (AGAf)
* Women with pregnancies complicated solely by early fetal growth restriction (before 34 weeks)
* Women with pregnancies complicated solely by late fetal growth restriction (after 34 weeks)
* Women identified as high-risk in first-trimester screening for preeclampsia Women identified as high-risk in first-trimester screening for fetal growth restriction
* Low-risk pregnancies in first-trimester screening for preeclampsia and fetal growth restriction, with physiological follow-up visits until delivery (homogeneous control sample)

Exclusion Criteria:

* Multiple pregnancies
* Pregnancies complicated by major fetal abnormalities identified during the 11-13 week gestational assessment
* Women who are unconscious or severely ill, women with learning difficulties, and those with severe psychiatric disorders
* Age <18 years
* Women who have not provided informed consent for the study
* Women with HIV, HBV, HCV infection
* Women with a history of leukemia and lymphoma
* Women with immunodeficiency
* Women who have used corticosteroids or other immunosuppressants in the last 3 months

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Women with pregnancies complicated by hypertensive disorders associated with or without fetal growth restriction in the second and third trimesters, and women identified as high-risk for the development of preeclampsia from the first trimester of pregnancy, will be offered the opportunity to participate in the study.
  To obtain a control sample, equal participation (1:1 ratio) of pregnant women identified as low-risk in first-trimester screening for preeclampsia and fetal growth restriction, who will undergo physiological follow-up visits until delivery, will also be requested. Recruitment of controls will follow an alternating principle: high risk-low risk-high risk-low risk.
  Patients will be followed up at defined intervals, varying depending on the underlying condition. High-risk patients and controls will be seen once per trimester if the pregnancy remains uncomplicated.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-06 (Actual); Primary Completion 2025-06-06 (Estimated); Study Completion 2025-06-06 (Estimated)

PRIMARY OUTCOMES:
Study of the Characteristics of Maternal Gut Microbiota in Women with Pregnancies Complicated by Hypertensive Disorders, with or without Fetal Growth Restriction. | through study completion, an average of 1 year
  Study of the characteristics of the microbiota in fecal samples from women with pregnancies complicated by hypertensive disorders, with or without fetal growth restriction.
Study of the Characteristics of Metabolome, in Women with Pregnancies Complicated by Hypertensive Disorders, with or without Fetal Growth Restriction. | through study completion, an average of 1 year
  Study of the characteristics of the metabolites in fecal and blood samples from women with pregnancies complicated by hypertensive disorders, with or without fetal growth restriction.
Study of the Characteristics of NK and B Cells in Women with Pregnancies Complicated by Hypertensive Disorders, with or without Fetal Growth Restriction. | through study completion, an average of 1 year
  Study of the characteristics of NK and B cells in blood samples from women with pregnancies complicated by hypertensive disorders, with or without fetal growth restriction.

SECONDARY OUTCOMES:
Study of the Characteristics of Microbiota in Women with Pregnancies | through study completion, an average of 1 year
  Assessment of Changes in Maternal Microbiota, in High-Risk Patients in the First Trimester for Preeclampsia or Fetal Growth Restriction
Study of the Evolution of Metabolome in Women with Pregnancies | through study completion, an average of 1 year
  Assessment of Changes in Maternal Metabolites in High-Risk Patients in the First Trimester for Preeclampsia or Fetal Growth Restriction
Study of the Evolution of NK and B Cells in Women with Pregnancies | through study completion, an average of 1 year
  Assessment of Changes in B and NK Cells in High-Risk Patients in the First Trimester for Preeclampsia or Fetal Growth Restriction
Evaluation of a Possible Correlation Between Dietary Habits and Maternal Gut Microbiota | through study completion, an average of 1 year
  The diet record will be obtained through a validated questionnaire on dietary habits and lifestyle. Spearman correlation of α-diversity microbiota measures and dietary intake will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas University, Pieve Emanuele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided